CLINICAL TRIAL: NCT01499914
Title: Cohort Study Evaluating the Clinical Effectiveness, Safety and Immunogenicity to the Pandemic Influenza Vaccination in Patients With Cystic Fibrosis and, Where Applicable, the Clinical Expression of Influenza A (H1N1)
Brief Title: Cohort Study Evaluating the Clinical Effectiveness, Safety and Immunogenicity to the Pandemic Influenza Vaccination
Acronym: MUCOFLU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P 100201; 2009-016662-90 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-12-26 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis With Gastrointestinal Manifestation
Keywords: vaccination H1N1; cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Influenza vaccination (Experimental): Influenza vaccination in patients with cystic fibrosis
  Interventions: Biological: influenza vaccination

INTERVENTIONS:
Biological: influenza vaccination — Influenza vaccination in patients with cystic fibrosis

SUMMARY:
Multicenter prospective cohort of approximately 1000 cystic fibrosis patients followed in the Ile de France during the 2009-2010 influenza season with the main objective to assess the effectiveness of antiviral vaccination (H1N1). All subjects will be included, without excluding factor. In particular populations at risk are additional infants 6 to 23 months, pregnant women and lung transplant will also be included. These people will be vaccinated with un-adjuvanted vaccine.

If flu symptoms until the results of PCR to confirm or refute the diagnosis of influenza, oseltamivir is administered in accordance with official recommendations and based on the results of the pharmacokinetic study.

DETAILED DESCRIPTION:
Main objective : To investigate the clinical efficacy of pandemic influenza vaccine (H1N1) v patients with cystic fibrosis (CF)

Secondary objectives : Vaccine research

* Measure the adherence of this population to the pandemic influenza vaccination
* Measure the tolerance of the pandemic influenza vaccine (H1N1) v
* Study the immunogenicity vaccine against the H1N1 variant and factors associated with vaccine response

Epidemiological and clinical study :

* Describe the incidence of asymptomatic forms of influenza A (H1N1) among unvaccinated and identify factors associated with the occurrence of these forms in patients with cystic fibrosis
* Describe the impact of influenza A (H1N1) in vaccinated and unvaccinated
* Characterizing the clinical expression of the influenza pandemic period in vaccinated and unvaccinated and identify factors associated with the occurrence of severe forms in patients with cystic fibrosis
* Characterize the serological response in patients who have a proven H1N1
* Characterize the impact of influenza A (H1N1) on the lung disease patients in the short and medium term

Virological study :

* Description of the epidemiology of respiratory viruses and intracellular bacteria involved in influenza-like illness
* In-context of H1N1 infection:
* Study of co-infections by intracellular bacteria or viral
* Quantification of viral RNA in respiratory secretions
* Monitoring the kinetics of viral shedding and correlation of it to the severity of respiratory disease and immunological protection
* Sensitivity analysis of viral strains to antiviral drugs and search for potential selection of resistant strains in antiviral therapy

Genomic study :

Search for susceptibility genes increase the risk:

* A severe form
* A prolonged viral shedding (beyond day 10), including research polymorphism carboxylesterase 1
* A immunoprotection

Methodology :

Prospective, multicenter, nonrandomized. Multicenter prospective cohort of approximately 1000 CF patients followed in the Ile de France during the 2009-2010 influenza season

* All patients with CF followed in Ile de France and the two transplant centers (IDF service of Thoracic Surgery at the European Hospital Georges Pompidou and Foch) will be included as much as possible, about 1000 patients (about 600 children).
* 200 of them (100 children at least 6 months, 100 adults) participate in the study of immunogenicity after vaccination
* 6 patients over 12 years will realize the pharmacokinetic study

Product under consideration :

Influenza vaccine (H1N1) v pandemic will be administered. It will mainly adjuvanted vaccine but also the un-adjuvanted vaccine in subjects at risk: infants 6 to 23 months, pregnant women, transplant.

If flu symptoms until the results of PCR to confirm or refute the diagnosis of influenza, oseltamivir is administered in accordance with official recommendations and based on the results of the pharmacokinetic study.

Criteria :

Primary endpoint :vaccine efficacy

To determine vaccine efficacy VE on susceptibility, the measure used is the complement to 1 of the Hazard Ratio (HR hazard ratio) for the appearance of an influenza episode (Halloran, AJE, 1997). The existence of an effective vaccine will be tested by comparing HR 1. Using the HR measurement is preferred to that using the ratio of cumulative incidence rates among vaccinated than unvaccinated because of a change in the number of groups vaccinated / unvaccinated can occur over time.

Indeed, the immunization schedule now includes two doses given at 3 weeks / 1 month apart, even if it appears that the antibody response can be achieved in the first half after the first dose. It is possible that some subjects may be infected before the first dose after the first but before the second, or after receiving the full presentation. On the other hand, the date of infection could be similar to that of vaccination, a time when efficiency is not optimal.

In the primary analysis, individuals will be considered unvaccinated if they do not receive vaccination and during 15 days of initial vaccination. For the latter, a time-dependent variable representing the immunization status will take into account their relative contribution to periods vaccinated / unvaccinated. The analysis will be stratified by age groups corresponding to the quartiles of the population.

In secondary analysis, the investigators vary the initial term conferring protection, the investigators also consider only those who received the full vaccination schedule, it will also determine the impact of using the cumulative incidence rate in the vaccinated population initially and ultimately vaccinated.

Secondary endpoints:

Membership in the vaccination will be measured as a proportion, together with a confidence interval 95%, as well as the incidence of clinical influenza in vaccinated and unvaccinated cohorts.

The tolerance of pandemic influenza vaccine (H1N1) v will be evaluated by binomial confidence intervals. Individual factors leading to the decision of vaccination and immunization events will be determined by logistic regression.

The clinical expression is described by the percentages of symptom onset. An analysis of the frequency of symptoms in groups of vaccination will be carried out. Factors related to the presence of symptoms will be sought using logistic regression. The percentage of serious forms will be measured. Vaccine efficacy against serious will be measured using techniques described by causal analysis Hudgens & Halloran.

The longitudinal lung function of patients enrolled will be analyzed through the data provided in the patient tracking software in place in services. A mixed effects linear model will be used to analyze changes in respiratory function (including FEV) and test whether the infection is accompanied by a change in the current level of functioning or a change in the evolution Compared to the situation pre-infection.

The pan-genomic analysis will evaluate SNPs (Single Nucleotide Polymorphisms) associated with the presence of (1) a prolonged infection, (2) of immunoprotection, (3) infection, (4) of a severe infection. Some patients, corresponding to extreme forms of the disease (severe and not severe) has been genotyped, and the whole cohort will be genotyped at term. Each patient has been genotyped about 300,000 SNPs. It is generally accepted that an association in this case is "genomically significant" when the significance level is smaller than 10-7. Actual calculations made in the project analysis of modifier genes Pr Clément, which resulted in the cohort, showed that in the comparison of two cohorts of 500 subjects, it was possible to obtain a significant result genomically a difference of about 20% between frequencies of genotypes for SNPs not rare (> 5%), with a risk factor (FDR) of approximately 10%. For the analysis of two groups of 150 subjects, under the same conditions, the FDR, however, was close to 1. The staff here will be compared between the two terminals, and often unbalanced. It is hoped to highlight the differences in genotype frequency, if any, of the order of 20% or more, in the case of a comparison involving the entire cohort, but the investigators will probably find that imbalances are larger (> 50%) in the analysis of smaller subgroups. In any case, it will be important to try and validate this information through independent study.

ELIGIBILITY:
Inclusion Criteria:

* patients with cystic fibrosis

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
immunogenicity of a A(H1N1)v influenza vaccine, administered in patients with cystic fibrosis | Day 21 for patients vaccinated with one dose of vaccine or Day 42 for patients vaccinated with 2 doses
  Immunogénicity was evaluated as:
  Seroprotection rate (defined by the percentage of patients with serum anti-haemagglutinin antibody titre ≥ 1/40e), seroconversion rate (defined by the percentage of patients with antibody titre <1/10e before vaccination and ≥ 1/40e after vaccination or with a titre ≥ 1/10e before vaccination and a titre at least 4-fold greater after vaccination) and seroconversion factor (defined by the ratio of the post/pre vaccination geometric mean titres) tested 3 weeks after the last influenza vaccination

SECONDARY OUTCOMES:
Vaccination tolerance: pain, erythema, fever, other general reactions | 1 year after vaccination
  Vaccination tolerance will be verified during all the study period
Longitudinal lung function evaluation, as asses | Before and 1 year after the day of vaccination
  FEV1, FVC recordings before and one year after the day of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Sermet, MD, PhD, Principal Investigator — Necker Hospital
Locations (1):
- Necker Hospital, Paris, France

REFERENCES:
- [Result] d'Alessandro E, Hubert D, Launay O, Bassinet L, Lortholary O, Jaffre Y, Sermet-Gaudelus I. Determinants of refusal of A/H1N1 pandemic vaccination in a high risk population: a qualitative approach. PLoS One. 2012;7(4):e34054. doi: 10.1371/journal.pone.0034054. Epub 2012 Apr 10. PMID 22506011
- [Result] Launay O, Boelle PY, Krivine A, Grenet D, Boussaud V, Remus N, Corvol H, Chedevergne F, Hubert D, Sermet-Gaudelus I; Inserm MUCOFLU group. Factors associated with humoral immune response to pandemic A/H1N1(v) 2009 influenza vaccine in cystic fibrosis. Vaccine. 2014 Jul 31;32(35):4515-4521. doi: 10.1016/j.vaccine.2014.06.010. Epub 2014 Jun 17. PMID 24950362
- [Derived] Bucher J, Boelle PY, Hubert D, Lebourgeois M, Stremler N, Durieu I, Bremont F, Deneuville E, Delaisi B, Corvol H, Bassinet L, Grenet D, Remus N, Vodoff MV, Boussaud V, Troussier F, Leruez-Ville M, Treluyer JM, Launay O, Sermet-Gaudelus I. Lessons from a French collaborative case-control study in cystic fibrosis patients during the 2009 A/H1N1 influenza pandemy. BMC Infect Dis. 2016 Feb 1;16:55. doi: 10.1186/s12879-016-1352-2. PMID 26830335